CLINICAL TRIAL: NCT04802798
Title: Gut Microbial Profiles in Fermentable Carbohydrate Induced Bloating: an Exploratory Double-blind, Randomized Cross-over, Trial
Brief Title: Pre-FIBRe Study: Predeterminants of Fibre Induced Bloating Response.
Acronym: Pre-FIBRe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Danone Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HR-19/20-18704
Record Dates: First submitted 2021-02-05; First posted 2021-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-01

CONDITIONS: Functional Bloating (Disorder)

STUDY DESIGN:
Intervention Model Description: cross-over study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo, Fibre 1, Fibre 2 (Experimental): All three interventions will be provided in a randomized double-blind order. The interventions will consist of 8 grams per day of three different types of powdered food supplement that will be mixed with water and consumed for a 7-day period. The powdered food supplement will be either placebo (glucose), fibre 1 (derived from a plant-based food) or fibre 2 (derived from a different plant-based food).
  Interventions: Dietary Supplement: Fibre 1; Dietary Supplement: Fibre 2; Dietary Supplement: Placebo
- Placebo, Fibre 2, Fibre 1 (Experimental): All three interventions will be provided in a randomized double-blind order. The interventions will consist of 8 grams per day of three different types of powdered food supplement that will be mixed with water and consumed for a 7-day period. The powdered food supplement will be either placebo (glucose), fibre 1 (derived from a plant-based food) or fibre 2 (derived from a different plant-based food).
  Interventions: Dietary Supplement: Fibre 1; Dietary Supplement: Fibre 2; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fibre 1 — Food derived fibre presented as a white powder
Dietary Supplement: Fibre 2 — Food derived fibre presented as a white powder
Dietary Supplement: Placebo — Simple sugar, presented as a white powder

SUMMARY:
This study is an exploratory study aimed at gaining a greater understanding of the cause of abdominal bloating in response to two distinct fibre types. This is a single-center, interventional double blinded randomized cross-over study. Each participant will consume each of the study products (placebo, fibre 1 and fibre 2) for a 7-day period with a 3-week washout period in between. Outcomes will be measured before and after each intervention period.

DETAILED DESCRIPTION:
The investigators have 4 hypotheses linked to 4 research questions that will be answered by this research:

Hypothesis 1: participants with self-reported functional bloating in response to either fibre-1 or fibre-2, but not both, will respond symptomatically to fibre-1 or fibre-2, defined as 'fibre-1 responders' and 'fibre-2 responders'.

Hypothesis 2: participants with functional bloating who are 'fibre-1 responders' will be distinguishable from 'fibre-1 non-responders', and 'fibre-2 responders' will be distinguishable from 'fibre-2 non-responders', based upon faecal microbial profiles identified using faecal metagenomics, transcriptomics and metabolites at baseline and following the fibre-1 and fibre-2 interventions.

Hypothesis 3: the microbiota, clinical and nutritional profiles of participants with functional bloating will be interrelated and these relationships will be distinguishable between 'fibre-1 responders', 'fibre-1 non-responders', and 'fibre-2 responders' and 'fibre-2 non-responders'.

Hypothesis 4: participants with visceral hypersensitivity will have different faecal microbiota and will be more likely to be a 'fibre-1 responders' or 'fibre-2 responders' than 'non-responders'.

Participants in the trial will take three different dietary substances, each at a dose of 8 grams per day (split into two serves of 4 gram doses) for 7-days in a double-blinded randomised order with a 3-week washout period in between each intervention. The products are provided in powdered format and will be mixed with water before drinking. The products being provided are glucose, and fibre-1 or fibre-2 (all extracts of commonly consumed food products).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults (18-60 years of age inclusive, and BMI 19-29 kg/m2 inclusive) who fulfil criteria for functional bloating as per Rome IV Criteria (to be assessed at screening phone call).
2. Individuals willing to provide consent and follow the protocol
3. Individuals who report that due to perceived trigger food avoidance, symptoms are well controlled i.e. report that over the past 3 days they have had absent or mild bloating on ≥2 days.
4. Individuals that do not fulfil Rome IV criteria for irritable bowel syndrome, functional constipation or functional diarrhoea
5. Individuals that report heightened bloating in response to foods predominantly high in just one type of study fibre i.e not those that report bloating in response to foods high in both. The goal will be to recruit equal proportion of each.
6. Individuals that are not diagnosed with any other chronic gastrointestinal disease or condition including inflammatory bowel disease, coeliac disease.

Exclusion Criteria:

* 1. Excessive habitual intake of fructans, galacto-oligosaccharides, polyols or fructose, as defined by clinician as the sole cause of symptoms.

  2. Individuals with specific diets (eg: strict low-FODMAP). 3. Participation in another clinical trial within the past 4 weeks 4. Subject with known or suspected allergy to any component of the study product(s).

  5. Individuals receiving treatment for anorexia, weight loss, or any form of treatment likely to interfere with metabolism or dietary habits.

  6. Vulnerable subjects defined as individuals whose willingness to volunteer in the clinical trial may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate. (Examples are members of a group with a hierarchical structure linked to the Investigator or to the Sponsor, such as students, subordinate hospital and laboratory personnel, employees of the Investigator or of the Sponsor).

  7. Individuals with antibiotics or proton pump inhibitor (e.g. omeprazole, lansoprazole and esomeprazole, pantoprazole, Rabeprazole) use within the previous 2 months 8. Individuals with current use of medication with potential central nervous system effects as judged by the investigator.

  9. Individuals with previous digestive surgery (except for appendectomy and cholecystectomy performed more than 2 years ago).

  10. Athletes as defined as performing daily strenuous daily exercise for more than 1.5 hours at a time.

  11. Oral disease that may impact on breath sampling e.g. gingivitis, halitosis, oral thrush, candidiasis.

  12. Individuals starting or routinely taking drugs (occasional use is acceptable) that might modify gastrointestinal function such as:
* Prokinetic agents e.g. metoclopramide (Reglan), tegaserod (Zelnorm), domperidone (Motilium),
* Anti-emetics agents
* Corticosteroids
* Narcotic analgesic agents e.g. methadone, fentanyl
* Anticholinergic agents for irritable bowel syndrome
* Medications for constipation e.g. enemas, cathartics, polyethylene glycol solutions, and lactulose.
* 5HT3 antagonists e.g. alosetron and ondansetron.
* Anti-diarrheal agents e.g. Imodium (loperamide)
* Opiate agents used to treat diarrhoea.
* NSAIDs e.g. ibuprofen
* Histamine2 blockers e.g. cimetidine (Tagamet), famotidine (Pepcid), and ranitidine hydrochloride (Zantac), nizatidine (Axid)
* Antacids e.g. Gaviscon, Maalox, Tums, or any that contain magnesium or aluminium
* Supplements used to treat bloating: activated charcoal, alpha galactosidase 13. Women who report they are pregnant/lactating/planning pregnancy 14. Recent/ongoing consumption of probiotics/prebiotic supplements (past 4 weeks) 15. Anticipated changes to consumption of naturally probiotic/prebiotic containing foods e.g. yogurt with live cultures or cereals with chicory etc, in the next 2 months 16. Anticipated changes to smoking habits in the next 2 months 17. Ongoing abuse of alcohol (>40 units per week)/non-prescription drugs/other medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Bloating as measured by the Gastrointestinal Symptom Rating Scale (GSRS) (Primary clinical response): end of first intervention period (day 7) | Day 7
  As this is an exploratory study to determine the underlying mechanisms of bloating the investigators have identified a primary and secondary symptom responder definition (those that become bloated in response to the intervention) that will be used to examine and compare the research outcome measures.
  The primary responder definition is: reporting moderate or severe bloating (a score of 2 or 3) on at least two of the final three days of the fibre-1 or fibre-2 challenge, measured using the Gastrointestinal Symptoms Rating Scale (GSRS), which rates individual gastrointestinal symptoms on a 4-point Likert scale (0-3). The primary responder definition of response will also be measured at the end of the placebo period.
Bloating as measured by the Gastrointestinal Symptom Rating Scale (GSRS) (Primary clinical response): end of second intervention period (day 35) | Day 35
  As this is an exploratory study to determine the underlying mechanisms of bloating the investigators have identified a primary and secondary symptom responder definition (those that become bloated in response to the intervention) that will be used to examine and compare the research outcome measures.
  The primary responder definition is: reporting moderate or severe bloating (a score of 2 or 3) on at least two of the final three days of the fibre-1 or fibre-2 challenge, measured using the Gastrointestinal Symptoms Rating Scale (GSRS), which rates individual gastrointestinal symptoms on a 4-point Likert scale (0-3). The primary responder definition of response will also be measured at the end of the placebo period.
Bloating as measured by the Gastrointestinal Symptom Rating Scale (GSRS) (Primary clinical response): end of third intervention period (day 63) | Day 63
  As this is an exploratory study to determine the underlying mechanisms of bloating the investigators have identified a primary and secondary symptom responder definition (those that become bloated in response to the intervention) that will be used to examine and compare the research outcome measures.
  The primary responder definition is: reporting moderate or severe bloating (a score of 2 or 3) on at least two of the final three days of the fibre-1 or fibre-2 challenge, measured using the Gastrointestinal Symptoms Rating Scale (GSRS), which rates individual gastrointestinal symptoms on a 4-point Likert scale (0-3). The primary responder definition of response will also be measured at the end of the placebo period.

SECONDARY OUTCOMES:
Secondary response measure: Adequate relief of bloating symptoms assessed by the Global Symptom Questionnaire (GSQ) (Secondary clinical response) | Day 7, day 21, day 28, day 35, day 56, day 63
  As this is an exploratory study to determine the underlying mechanisms of bloating the investigators have identified a primary and secondary clinical symptom responder definition (those that become bloated in response to the intervention) that will be used to examine and compare the research outcome measures.
  The secondary responder definition is: reporting not having adequate relief of bloating symptoms on at least two of the final three days of the fibre-1 or fibre-2 challenge, measured using the dichotomous Global Symptom Questionnaire (GSQ). The secondary responder definition of response will also be measured at the end of the placebo period.
Clinical profile: Gas-related gastrointestinal symptom profile assessed by the Intestinal Gas Questionnaire (IGQ) | Gas-related gastrointestinal symptom profile will be assessed after each intervention period (days 7, 35 and 63) and after each washout period (days 28 and 56) and once at a control timepoint (day 21).
  The IGQ is a multi-choice questionnaire that assesses 17 symptoms associated with abdominal gas production using a Likert scale (0-10).
Clinical profile: Gastrointestinal symptom profile assessed by the Gastrointestinal symptom rating scale (GSRS) | Gastrointestinal symptoms profile will be assessed after each intervention period (days 7, 35 and 63) and after each washout period (days 28 and 56) and once at a control timepoint (day 21).
  The GSRS is a 4-point Likert scale (0-3, absent-severe) assessing 16 gastrointestinal symptoms.
Clinical profile: Stool form and frequency using the Bristol Stool Form Scale (BSFS) | The BSFS for each stool passed will be recorded in a 7-day diary and will be assessed after each intervention period (days 7, 35 and 63) and after each washout period (days 28 and 56) and once at a control timepoint (day 21).
  The BSFS is a visual aid to help track stool form, stool form is ranked from type 1-7 and each stool passed will be recorded according to this scale.
Clinical profile: Abdominal girth (cms) | Abdominal girth will be recorded daily in a 7-day diary and will be assessed after each intervention period (days 7, 35 and 63) and after each washout period (days 28 and 56) and once at a control timepoint (day 21).
  Abdominal girth will be recorded daily using a visual guide for where to measure and a metric measuring tape.
Clinical profile: Visceral hypersensitivity - rectal barostat | Visceral hypersensitivity will be measured during the first washout period (between day 7 and day 28)
  Visceral hypersensitivity will be measured using a rectal barostat to measure rectal pressure tolerance (mm Hg) and provide a dichotomous hypersensitivity outcome (yes/no).
Nutrition profile: Energy and nutrient intake | Energy and nutrient intake will be recorded daily in a 7-day diary and will be assessed after each intervention period (days 7, 35 and 63) and after each washout period (days 28 and 56) and once at a control timepoint (day 21).
  Energy and nutrient analysis will be recorded in prospective 7-day diaries and assessed using computerised software (Nutritics) based on food composition data from standard United Kingdom (McCance and Widdowson 2016) food composition tables);
Nutrition profile: Fermentable oligo-, di-, mono- saccharide and polyol (FODMAP) intake | Dietary intake will be recorded daily in a 7-day diary and will be assessed after each intervention period (days 7, 35 and 63) and after each washout period (days 28 and 56) and once at a control timepoint (day 21).
  Diet diaries will be analysed for FODMAP intake using the Monash University FODMAP calculator.
Microbiome profile: Faecal transcriptomics from stool sample (microbiota activity) (metatranscriptomics profiling) | Days 21, 28, 35, 56, and 63
Microbiome profile: Faecal Volatile Organic Compounds (VOC) (gas-chromatography mass-spectrometry) from stool sample | Days 21, 28, 35, 56, and 63
Microbiome profile: Faecal Short-Chain Fatty Acids (SCFA) (gas-liquid chromatography) from stool sample | Days 21, 28, 35, 56, and 63
Microbiome profile: Fermentation (direct breath hydrogen and methane tests) using Gastrogenius breath-gas analyser | Days 21, 28, 35, 56, and 63

OTHER OUTCOMES:
Exploratory analysis of secondary outcome measures 5-15 (listed above) | Days 7, 21, 28, 35, 56, and 63
  Clinical, nutrition and microbiota profiles will be compared by further separating participants into four groups:
  fibre-1 only responders; fibre-2 only responders; responders to both challenges; responders to neither challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Whelan, PhD, Study Chair — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No